CLINICAL TRIAL: NCT04319913
Title: Whether Intraoperative Analgesia Guided by the Analgesia Nociception Index (ANI) Can Decrease the Amount of Narcotics, Other Anesthetic Drugs, and Blood Loss in Patients Undergoing Low-pressure Anesthesia: a Randomized Controlled Trial
Brief Title: ANI-guided Intraoperative Analgesia in Low-pressure Anesthesia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mackay Memorial Hospital (Other)
Responsible Party: Principal Investigator, Chien-Chung,Huang, Attending physician of anesthesiology , Principal Investigator, Mackay Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20MMHIS069e
Record Dates: First submitted 2020-03-20; First posted 2020-03-24 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Analgesia; Functional Endoscopic Sinus Surgery; Heart Rate Variability; Opioid Consumption
Keywords: analgesia nociception index; functional endoscopic sinus surgery; analgesia; opioid consumption; heart rate variability; low pressure anesthesia
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The analgesia nociception index sensors are a pair of patches. They would be placed on the participant's right shoulder and the left side of the chest before the induction of general anesthesia, recording the ANI value throughout the operation. In the control group, the ANI monitor would be covered up, so that the care provider could only titrate remifentanil based on clinical experience. The participants would be masked from which group they were allocated into. The surgeon would be masked from the participant's allocation, and surgeon's satisfaction to the operation field would be surveyed by a questionnaire right after the operation, also the estimated blood loss amount would be recorded by the same surgeon.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ANI-guided (Experimental): ANI-guided narcotics use to maintain ANI value between 50 to 70
  Interventions: Device: analgesia nociception index
- Control (No Intervention): narcotics use guided by clinical experience, ANI is still recorded but would be covered up intraoperatively

INTERVENTIONS:
Device: analgesia nociception index — Analgesia nociception index (ANI) could objectively monitor how pain the participant is. In the experimental group, the care provider would decrease the dose of narcotics (remifentanil) if the ANI value is above 70, and increase the dose if the ANI value is under 50.
  Arms: ANI-guided

SUMMARY:
During functional endoscopic sinus surgery(FESS), low-pressure anesthesia is often applied, aiming to decreased operative blood loss, and anesthetics, narcotics and antihypertensive agents are given to achieve desirable low blood pressure. However, the dose of these medications given is usually decided subjectively based on the clinical experience of the care provider, placing the patient in a risky situation of narcotics overdosing or underdosing. Therefore, here is the question: Whether intraoperative analgesia guided by an objective pain monitoring device, such as the Analgesia Nociception Index (ANI), could decrease the amount of narcotics, other anesthetic agents, and blood loss in patients undergoing low-pressure anesthesia.

DETAILED DESCRIPTION:
Analgesia nociception index (ANI) is an objective pain monitoring device, it could measure parasympathetic tone base on heart rate variability analysis, which is a way to measure the effect of respiratory sinus arrhythmia on heart rate. In the previous studies, ANI had been used to predict immediate postoperative pain, intraoperative analgesia in children, and intraoperative analgesia in bariatric surgery, which showed ANI can be used to detect surgical stimuli, reduce intraoperative consumption of narcotics, and assess immediate postoperative pain intensity. However, no publication has mentioned ANI been used in low-pressure anesthesia.

Participants with ASA physical status class I or II, age between 20-65, and body mass index less than 35 who would undergo FESS are enrolled and randomly allocated by using computer-generated random number table into two groups with equal probability: ANI-guided remifentanil titration or remifentanil titration by standard care. Total intravenous anesthesia with propofol TCI(target controlled infusion) and remifentanil TCI are used for anesthesia maintenance, targeting bispectral index between 40 and 60. The ANI value in experimental group would be maintained between 50 and 70. Intraoperative mean arterial pressure (MAP) would be targeted at 55-65 mmHg, and calcium channel blocker would be administered if MAP could not achieve target despite of propofol and remifentanil titration.

Participant's demographics, baseline information, type and duration of the operation, duration from end of the surgery till participant awaken, ANI value, vital signs, the amount of narcotics, anesthetics and antihypertensive medications used, intraoperative blood loss, surgeon's satisfaction to the operation field, participant first recorded pain score in postoperative recovery room using visual analogue scale, and opioid-associated side effects such as nausea, vomiting, pruritis, dizziness in postoperative recovery room, will be recorded and analyzed. The statisticians will apply Chi-square for categorical data, T-test for continuous data, and multiple regressions analysis. P value less than 0.05 was considered statistically significant. Using G-power software to estimate, predicted sample size is 120 presuming type I error 0.05, power 0.95, and medium effect size.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status class I or II
* age between 20-65
* body mass index less than 35
* scheduled for functional endoscopic sinus surgery

Exclusion Criteria:

* major cardiovascular disease, arrhythmia, respiratory disease, cerebral vascular disease, or ASA physical status classification III or greater
* documented or self-reported history of chronic pain
* acute or chronic opioid analgesic use
* dysautonomia
* diabetes mellitus with evidence of neuropathy
* emergency cases
* allergy to medications in the study

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Narcotics consumption | From the first given dose of remifentanil until the last given given dose of remifentanil during anesthesia, assessed up to 8 hours.
  Remifentanil would be used as narcotics, the total amount used intraoperatively would be recorded

SECONDARY OUTCOMES:
Anesthetics consumption | From the first given dose of anesthetics (propofol or midazolam, whichever comes first) until the last given given dose of anesthetics (propofol or midazolam, whichever comes last), assessed up to 8 hours.
  The amount of anesthetics (mainly propofol) used intraoperatively would be recorded

OTHER OUTCOMES:
Blood loss | the estimated blood loss would be recorded immediately after the operation
  Blood loss would be estimated by surgeon
Bleeding of the operation field | The questionnaire would be provided to the surgeon immediately after the operation
  Bleeding of the operation field would be surveyed to surgeons by a questionnaire.
  The clarity of operation field:
  1. Minimal bleeding: no need of suction.
  2. Slightly bleeding: suction sometimes.
  3. Moderate bleeding: Suction frequently
  4. Severe bleeding: surgical field compromised even right after suction
  5. Continuous bleeding.

CONTACTS AND LOCATIONS:
Overall Officials: Chien-Chung Huang, MD, Study Director — Mackay Memorial Hospital
Locations (1):
- MacKay Memorial Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Boselli E, Bouvet L, Begou G, Dabouz R, Davidson J, Deloste JY, Rahali N, Zadam A, Allaouchiche B. Prediction of immediate postoperative pain using the analgesia/nociception index: a prospective observational study. Br J Anaesth. 2014 Apr;112(4):715-21. doi: 10.1093/bja/aet407. Epub 2013 Dec 8. PMID 24322571
- [Background] Julien-Marsollier F, Rachdi K, Caballero MJ, Ayanmanesh F, Vacher T, Horlin AL, Skhiri A, Brasher C, Michelet D, Dahmani S. Evaluation of the analgesia nociception index for monitoring intraoperative analgesia in children. Br J Anaesth. 2018 Aug;121(2):462-468. doi: 10.1016/j.bja.2018.03.034. Epub 2018 Jun 5. PMID 30032886
- [Background] Le Gall L, David A, Carles P, Leuillet S, Chastel B, Fleureau C, Dewitte A, Ouattara A. Benefits of intraoperative analgesia guided by the Analgesia Nociception Index (ANI) in bariatric surgery: An unmatched case-control study. Anaesth Crit Care Pain Med. 2019 Feb;38(1):35-39. doi: 10.1016/j.accpm.2017.09.004. Epub 2017 Oct 12. PMID 29033356